CLINICAL TRIAL: NCT04087252
Title: PhaseI Trial of Tumor Neoantigen Vaccine
Brief Title: An Immunogenic Personal Neoantigen Vaccine for Cancer Treatment
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HN2019NIP
Record Dates: First submitted 2019-09-03; First posted 2019-09-12 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2019-08

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- vaccinated group (Experimental): Neoantigen vaccination will be performed with 6 doses in total, once per week
  Interventions: Biological: tumor neoantigen

INTERVENTIONS:
Biological: tumor neoantigen — tumor neoantigens

SUMMARY:
Despite years of preclinical efforts and hundreds of clinical studies, therapeutic cancer vaccines with the routine ability to limit or eliminate tumor growth in humans have been elusive. With advances in genome sequencing, it is now possible to identify a new class of tumor-specific antigens derived from mutated proteins that are present only in the tumor. These "neoantigens" should provide highly specific targets for antitumor immunity. Although many challenges remain in producing and testing neoantigen-based vaccines customized for each patient, a neoantigen vaccine offers a promising new approach to induce highly focused antitumor T cells aimed at eradicating cancer cells

DETAILED DESCRIPTION:
1. Methods of vaccine storage and transportation: as a special biological product, the vaccine should be stored at 2-8 ℃ to protect the efficacy (titer) of the vaccine from being damaged.All vaccines must be stored and transported at temperatures that meet regulatory requirements.A cold chain system is required to support and monitor the temperature at all stages of the vaccine from production to final inoculation (aircraft, ship, train, automobile, motorcycle, bicycle, walking, etc.);Cold storage, refrigerator, vaccine transport box, cold pack, ice bar, etc.) to avoid overheating or over-cooling.
2. Treatment plan: intramuscular injection of vaccines of D1, D4, D7, D14, D21, D51, D142 of the deltoid muscle of the left and right upper arm, every six months for the next 3 years, and every year for the next 3 years, until the patient withdrew from the clinical study or the study was discontinued.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years ≤ 70 years at the time of informed consent
* Signed informed consent to be provided
* failed in previous standard chemotherapy and targeted therapy
* Life expectancy not less than 90 days
* Karnofsky performance status 0-1
* adequate organ functions

Exclusion Criteria:

* Actively infectious condition including hepatitis
* Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the treatment on the fetus or infant.
* Any form of primary immunodeficiency (such as Severe Combined immunodeficiency Disease).
* Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities).
* Active systemic infections, coagulation disorders or any other active major medical illnesses.
* Patients who are receiving any other investigational agents.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-09-04 (Actual); Primary Completion 2021-10-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety of the immunogenic personal neoantigen vaccine | 1.5 years
  The incidence of serious adverse events

SECONDARY OUTCOMES:
Disease control rate | 1 year
  It is defined as the proportion of complete response, partial response and stable disease

CONTACTS AND LOCATIONS:
Overall Officials: Ning Li, PhD, Principal Investigator — Henan Cancer Hospital; Suxia Luo, PhD, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China